CLINICAL TRIAL: NCT02403128
Title: Intravitreal Aflibercept Injection for Symptomatic Macular Edema From Retinal Artery Macroaneurysms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kamal Kishore, MD (Other)
Responsible Party: Sponsor-Investigator, Kamal Kishore, MD, Principal Investigator, Illinois Retina and Eye Associates
Organization: Illinois Retina and Eye Associates (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kishore_Eylea_RAM
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Macular Edema; Retinal Artery Macroaneurysm
Keywords: 362.17
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with macular edema from RAM (Experimental): Intravitreal aflibercept 2.0 mg injection for eyes meeting eligibility criteria will be administered at baseline. Reinjection of the drug for protocol-defined criteria at least two months after previous injection.
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — Intravitreal injection of 2.0 mg aflibercept at baseline, and repeated no sooner than two months from the previous injection for persistent macular edema as defined in the protocol.
  Other Names: Eylea

SUMMARY:
Phase 1, non-randomized, open label, noncomparative trial to study the effect of intravitreal injection of aflibercept on eyes with symptomatic macular edema from retinal artery macroaneurysms.

DETAILED DESCRIPTION:
Baseline evaluation will consist of measurement of best-corrected ETDRS visual acuity, complete eye exam, including IOP measurement, color photos and intravenous fluorescein angiography, spectral domain OCT and vitals. Patients meeting eligibility criteria will be treated with an intravitreal injection of 2.0 mg aflibercept under usual aseptic precautions. Follow up visits will be on Day 7, 30, 60, 90, 120, 150 and 180. At each follow-up visit, best-corrected ETDRS visual acuity, IOP measurement and central foveal thickness (CFT) by SDOCT will be obtained. Color photos and IVFA will be performed at month 3 and 6 visits.

Retreatment shall be performed no sooner than two months after previous injection for one or more the following criteria 1. CFT >310 microns 2. Intraretinal or subretinal fluid on SDOCT 3. Increase in CFT by 50 or more microns from the lowest value observed after intravitreal aflibercept injection 4. Decrease in vision by 5 or more letters frpm the previous visit associated with OCT evidence of macular edema. 5. Appearance of new hemorrhage on color photographs.

Final follow-up will be at six months. Data collected will include, change in ETDRS visual acuity from the baseline, change in CFT, number of injections, number of eyes completely dry by SDOCT, and number of eyes with a thrombosed RAM by IVFA.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic macular edema caused by RAM in one of the eyes. If both eyes are involved, the eye with worse central foveal thickness will be enrolled in the study.
2. CFT of 310 microns or more by spectral domain OCT or lipid in the center of the fovea
3. Best-corrected visual acuity of 73 to 24 letters.
4. Willing and able to comply with clinic visits and study-related procedures.
5. Willing to provide informed consent -

Exclusion Criteria:

1. Media opacity
2. pre-retinal fibrosis, retinal detachment, vitreo-macular traction
3. Infectious keratitis, conjunctivitis, blepharitis or scleritis
4. Any ocular surgery during the preceding 3 months.
5. aphakia or uncontrolled glaucoma
6. subfoveal hemorrhage
7. History of systemic or intravitreal anti-VEGF injections, intravitreal steroid injection or implant, or laser treatment to RAM within six months
8. Any other ocular disease responsible for decrease in vision.
9. Concomitant ocular disease that can cause increase in foveal thickness
10. Ocular inflammation from any cause
11. Recent (<3 months) history of a thromboembolic event
12. Pregnant or breast feeding women.
13. Sexually active men or women of child bearing potential who are unwilling to practice adequate contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Safety profile as demonstrated by the incidence and severity of ocular and systemic adverse events in patients with macular edema caused by retina artery macroaneurysm(s) after intravitreal injection of 2 mg of aflibercept | six months

SECONDARY OUTCOMES:
Change in best-corrected ETDRS visual acuity at 3 and 6 months. | six months.
Change in central field macular thickness at 3 and 6 months | six months
Proportion of eyes completely dry by spectral domain OCT | six months
Occlusion of retinal artery macroaneurysm (RAM) at 3 and 6 months by intravenous fluorescein angiography | six months
Number of patients requiring additional treatment beyond baseline and total number of treatments | six months

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Kishore, MD, Principal Investigator — Illinois Retina and Eye Associates
Locations (1):
- Illinois Retina and Eye Associates, Peoria, Illinois, United States